CLINICAL TRIAL: NCT04125979
Title: Clinical Application of Vagus Nerve Preservation in Minimally Invasive Surgery for Early Lung Cancer
Brief Title: Clinical Evaluation of Vagal Nerve Preservation in Minimally Invasive Surgery for Early Lung Cancer
Acronym: CEVNPIMISELC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Yongxin Zhou, Director, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-LCYJ-006
Record Dates: First submitted 2019-10-05; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer Stage I
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: 120 patients were divided into two groups. One group retained the pulmonary vagus nerve and the other group severed the vagus nerve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preservation of pulmonary vagus nerve (Experimental): Preservation of pulmonary branches of vagus nerve in minimally invasive surgery for lung cancer
  Interventions: Other: In minimally invasive surgery，Vagus nerve preservation
- No pulmonary vagus nerve preservation (Experimental): In minimally invasive surgery for lung cancer, the pulmonary branches of vagus nerve were severed
  Interventions: Other: In minimally invasive surgery，Vagus nerve is not preserved

INTERVENTIONS:
Other: In minimally invasive surgery，Vagus nerve preservation — In minimally invasive surgery for lung cancer, the experimental group retained the pulmonary branches of vagus nerve
  Arms: Preservation of pulmonary vagus nerve
Other: In minimally invasive surgery，Vagus nerve is not preserved — In minimally invasive surgery for lung cancer, the control group did not retain the vagus nerve.
  Arms: No pulmonary vagus nerve preservation

SUMMARY:
Through prospective, randomized and controlled clinical study, patients with early lung cancer who do not need lymph node dissection according to routine diagnosis and treatment were selected. The feasibility and safety of preserving vagal pulmonary branch intact during minimally invasive surgery were compared with traditional minimally invasive surgery, and the feasibility and safety of preserving vagal pulmonary branch intact during minimally invasive surgery were clarified. The effect of preserving pulmonary branches of vagus nerve in minimally invasive surgery of early lung cancer on preventing or reducing pulmonary complications after operation was evaluated by main observation indexes (incidence of pulmonary complications) and secondary evaluation indexes. It will provide a safer, simpler and more effective new technology for patients with early lung cancer undergoing minimally invasive surgery, and provide a basis for the popularization of this new technology.

DETAILED DESCRIPTION:
According to the suggestion of statistical experts and the minimum sample size, 120 IA1-2 patients who are going to undergo thoracoscopic lung surgery were selected according to the criteria of admission and exclusion. The risk and benefit were informed and the informed consent of the subjects was signed. The patients were numbered and randomly divided into two groups: group A with vagus nerve preservation during minimally invasive surgery and group B with traditional minimally invasive surgery for early lung cancer. The incidence of pulmonary complications within 5 weeks after operation (see the evaluation criteria for details), operation time, intraoperative bleeding volume, postoperative drainage volume, postoperative mortality, incidence of cardiovascular complications, rate of re-tracheal intubation, rate of re-admission to ICU, duration of stay in ICU, hospitalization costs were observed. Statistical analysis and evaluation of the safety of preserving pulmonary branches of vagus nerve in minimally invasive surgery and the effectiveness of preventing or reducing pulmonary complications after minimally invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18-70 years of age, regardless of gender;
* (2) From May 2019 to December 2021, patients with lung cancer who underwent thoracoscopic pneumonectomy (wedge-shaped, segment and lobe) were admitted to our hospital. Postoperative pathological diagnosis was non-small cell lung cancer. Preoperative pathological staging was T1a-bN0M0 and IA1-2 (pathological staging refers to UICC 8th Edition TNM staging standard for lung cancer).
* (3) In addition to routine examinations, all patients underwent enhanced chest CT, cranial CT/MRI, abdominal B-mode ultrasound, whole body bone isotope scan or PET-CT to exclude distant metastasis.
* (4) Subjects clearly understand the purpose of the study, are willing and able to comply with the requirements to complete the study, and sign the informed consent.

Exclusion Criteria:

* (1) Patients with other infectious diseases (inflammation, tuberculosis, etc.) in the thoracic cavity;
* (2) Patients are unwilling to accept the new technique of preserving pulmonary branch of vagus nerve during operation;
* (3) Clinical unstable patients with severe cardiovascular, renal and respiratory system;
* (4) Participated in other clinical trials within 30 days;
* (5) Other reasons why researchers think it is inappropriate to participate in the experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
cough after pulmonary resection | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  (1) dry cough lasting no less than 2 weeks after pneumonectomy; (2) no obvious abnormalities in chest X-ray; (3) excluding drug factors such as postnasal drip syndrome, bronchial asthma and ACEI
pulmonary infection | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Postoperative pneumonia should be considered if there are three or more of the following indicators:
  1. Fever occurred 72 hours after operation, and the body temperature increased again within T > 38 C or 72 hours.
  2. Leukocyte count increased (>12-15*109/L) or increased again after the leucocyte count returned to normal value, exceeding 10*109/L;
  3. Chest imaging showed consolidation of lung tissue or increasing patchy shadow;
  4. cough up purulent sputum or sputum culture positive;
  If it contains 4, only one of the other items can be considered as a respiratory consultation to determine pulmonary infection, and need to replace antibiotics or prolong the use of antibiotics.
Atelectasis | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  (1) Imaging findings suggest atelectasis or consolidation of the lungs; (2) signs of dyspnea; (3) decreased oxygen saturation to below 90%.
hydrothorax | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Re-catheterization was needed; dyspnea symptoms; and drainage time was longer than 15 days.
Postoperative respiratory failure or ARDS or requiring tracheal intubation | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Tracheal intubation; Ventilator; ICU

SECONDARY OUTCOMES:
Operation time; | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Operation time;
Intraoperative bleeding volume; | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Intraoperative bleeding volume;
Postoperative drainage volume; | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Postoperative drainage volume;
Postoperative mortality | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Postoperative mortality
Postoperative cardiovascular complications | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Postoperative cardiovascular complications
Re-admission ICU rate; | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Re-admission ICU rate;
Time of stay in ICU; | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Time of stay in ICU;
Hospitalization days | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Hospitalization days
Hospitalization expenses | From the date of randomized grouping to 5 weeks after operation, the evaluation time was as long as 5 weeks.
  Hospitalization expenses

CONTACTS AND LOCATIONS:
Overall Officials: Yongxin zhou, Doctor, Study Director — Tongji Hospital affiliated to Tongji University
Locations (1):
- Yongxin Zhou, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen W, Zheng R, Zeng H, Zhang S. Epidemiology of lung cancer in China. Thorac Cancer. 2015 Mar;6(2):209-15. doi: 10.1111/1759-7714.12169. Epub 2015 Mar 2. PMID 26273360
- [Result] Sawabata N, Maeda H, Takeda S, Inoue M, Koma M, Tokunaga T, Matsuda H. Persistent cough following pulmonary resection: observational and empiric study of possible causes. Ann Thorac Surg. 2005 Jan;79(1):289-93. doi: 10.1016/j.athoracsur.2004.06.045. PMID 15620960
- [Result] Sarna L, Evangelista L, Tashkin D, Padilla G, Holmes C, Brecht ML, Grannis F. Impact of respiratory symptoms and pulmonary function on quality of life of long-term survivors of non-small cell lung cancer. Chest. 2004 Feb;125(2):439-45. doi: 10.1378/chest.125.2.439. PMID 14769722
- [Result] Weijs TJ, Goense L, van Rossum PSN, Meijer GJ, van Lier AL, Wessels FJ, Braat MN, Lips IM, Ruurda JP, Cuesta MA, van Hillegersberg R, Bleys RL. The peri-esophageal connective tissue layers and related compartments: visualization by histology and magnetic resonance imaging. J Anat. 2017 Feb;230(2):262-271. doi: 10.1111/joa.12552. Epub 2016 Sep 23. PMID 27659172
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=2.%09Chen+W%2C+Zheng+R%2C+Zeng+H%2C+et+al.+Epidemiology+of+lung+cancer+in+China.+Thorac+Cancer%2C+2015%2C+6(2)%3A+209-215.
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/?term=Persistent+cough+following+pulmonary+resection%3A+observational+and+empiric+study+of+possible+causes
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/14769722
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=Theperi-esophageal+connective+tissue+layers+and+related+compartments%3A+visualization+by+histology+and+magnetic+resonance+imaging.